CLINICAL TRIAL: NCT01586559
Title: Evaluation of the Long-term Stability of Sheath Plication Using Absorbable Sutures in Patients With Diastasis of the Recti Muscles: an Ultrasonography Study
Status: Completed | Type: Observational
Sponsor: Bulovka Hospital (Other)
Responsible Party: Principal Investigator, Ondrej Mestak M.D., Ondrej Mestak M.D., Bulovka Hospital
Other Study IDs: IGANT11 392-6/2010-1
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Diastasis Recti

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Control group: Nulliparous women
- Diastasis: Patients after rectus sheath plication due to diastasis

SUMMARY:
A comparative prospective study assessing the outcomes of recti muscle diastasis correction with absorbable suture.

DETAILED DESCRIPTION:
Background: Rectus sheath plication within abdominoplasty is a standard treatment for diastasis of the recti muscles. Previous studies assessing the efficacy and endurance of the correction of recti diastasis have mostly been performed with small groups of patients, short follow-up periods and/or with questionable methodology

Methods: A comparative prospective study assessing the outcomes of recti muscle diastasis correction with absorbable suture. The investigators assess the outcomes by physical and ultrasonographic examinations and a patient questionnaire, which asks about the number of pregnancies and the types of deliveries, other abdominal surgeries before or after the abdominoplasty, the interval of time required to return to full activity, postoperative pain, and the overall satisfaction with the final result. During the examination, the inter-recti distances are measured at 3 levels: halfway between the xyphoid and umbilicus, just above the umbilicus and halfway between the umbilicus and pubis. The same examination is done on a control group of nulliparous women.

ELIGIBILITY:
Inclusion Criteria:

Women after rectus sheath plication for diastasis recti

Exclusion Criteria:

Abdominal wall defect other then umbilical hernia

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with interval after rectus sheath plication
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of the long-term stability of sheath plication using absorbable sutures in patients with diastasis of the recti muscles | 12-41 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bulovka Hospital, Prague, Czechia